CLINICAL TRIAL: NCT06239142
Title: Mental Fatigue and Outcome After Subarachnoid Hemorrhage
Brief Title: Understanding Mental Fatigue After Subarachnoid Hemorrhage
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Helena Odenstedt Hergès, Associate professor, Sahlgrenska University Hospital
Other Study IDs: SAH I
Record Dates: First submitted 2024-01-25; First posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Subarachnoid Hemorrhage, Aneurysmal; Mental Fatigue
MeSH Terms: conditions — Subarachnoid Hemorrhage; Mental Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Fatigue is among the most frequently reported sequelae in stroke survivors. For a specific stroke diagnosis, aneurysmal subarachnoid hemorrhage (aSAH), fatigue, in general, is reported to be present in 30 to 90% of the patients. It is the mental fatigue component that significantly contributes to difficulties that patients with aSAH face when returning to normal life. However, there is substantial variation in the reported incidence of mental fatigue (25%-60%), which may be attributed to several methodological factors, such as differences in the follow-up periods and instruments used. Consequently, a complete understanding of how mental fatigue influences long-term recovery remains elusive. This research project will contribute to new and important knowledge in long-term effects after SAH when it comes to mental fatigue.

In this study patients surviving an SAH will be assessed for mental fatigue at 5 years after the insult. The patients have previously been assessed at 1 and 3 years. All patients have been treated at Sahlgrenska University Hospital during the acute phase after SAH. Follow-up is performed after 5 years after aSAH through a structured telephone interview, where patients are scored using the Glasgow Outcome Scale-Extended (GOSE) Additionally, the patients receive a self-assessment questionnaire, the Mental Fatigue Scale, Patients are reminded to return the questionnaires at three times.

This study aims to determine the long-term prevalence, severity, and dynamics of mental fatigue at 1, 3, and 5 years after an aSAH. The study also aims to identify whether demographic characteristics and secondary complications or diagnoses after aSAH can be associated with an increased risk of developing mental fatigue or unfavourable outcome.

DETAILED DESCRIPTION:
In this study patients surviving an SAH will be assessed for mental fatigue at 5 years after the insult. The patients have previously been assessed at 1 and 3 years. All patients have been treated at Sahlgrenska University Hospital during the acute phase after SAH. Follow-up is performed after 5 years after aSAH through a structured telephone interview, where patients are scored using the Glasgow Outcome Scale-Extended (GOSE) Additionally, the patients receive a self-assessment questionnaire, the Mental Fatigue Scale, Patients are reminded to return the questionnaires at three times.

Primary outcome measure:

The Mental Fatigue Scale (MFS)score

The MFS is a multidimensional self-reporting questionnaire developed for assessing different aspects of mental fatigue in patients with brain injuries. It comprises 15 items regarding fatigue, including lack of initiative; mental recovery; concentration difficulties; memory problems; slowness of thinking; sensitivity to stress; increased mental fatigue, increased tendency to become emotional; irritability; sensitivity to light and noise; and decreased or increased sleep duration. Each item has four response options ranging from 0 (normal function) to 3 (maximal problems); further, one can select response points in between (i.e., 0,5, 1,5, and 2,5), which yields a total of seven options. Items 1-14 are used to calculate the total score, with a maximum score of 42. We did not include item 15, which assesses 24-h variations, in the total score, but it can be used in clinical practice. An MFS score ≥ 10.5 indicates mental fatigue. A higher MFS score indicates more severe problems.

This study explores the presence, severity and dynamics of mental fatigue.

The Glasgow Outcome Scale-Extended (GOSE)

The GOSE evaluates the patient's functional outcome and level of independence in eight different domains of daily living, including physical, cognitive, emotional, and social functioning. It was developed to classify patients after a traumatic or nontraumatic brain injury, allowing for comparisons of outcomes between patients. The scale ranges from death (1 point) to good recovery (8 points), with higher scores indicating better outcomes and higher levels of independence. A GOSE score of 8 indicates full recovery with only minor symptoms that do not affect activities of daily living (ADL). A GOSE score of ≥ 5 indicates that patients can independently manage their ADL and is used in studies to describe a favorable outcome 5,28.

Secondary Outcome Measures are the association between mental fatigue and GOSE, demographics, complications during the acute phase and loss of conscious at ictus.

ELIGIBILITY:
Inclusion Criteria:

* Patients having had a aneurysmal subarachnoid hemorrhage

Exclusion Criteria:

* age<18 years, patients having pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 64 patients where included in a primary study of the acute phase after subarachnoid hemorrhage. This study population consists of patients surviving up to 5 years after the SAB and eligible to assess for the presence of mental fatigue.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2021-10 (Actual); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Mental fatigue | 5 years
  Mental fatigue scale score. The instrument consists of 15 questions addressing different problems within the fatigue area and problems can be graded by the patient in 7 steps according to severity. Maximum score is 30 and a value above 10.5 indicates the presence of mental fatigue.
GOSE | 5 years
  extended Glascow outcome scale. Describing functional outcome according to an 8-grdaed scale where 1 corresponds to dead and 8 to fully recovered.

CONTACTS AND LOCATIONS:
Overall Officials: Helena Odenstedt Herges, PhD, Principal Investigator — Sahlgrenska Academy Gothenburg University Inst of Clinical sciences

IPD SHARING:
Plan to Share IPD: No
Individual patient data will not be shared